CLINICAL TRIAL: NCT02981017
Title: Prospective Study for Improvement in Outcomes Following Draf III/Endoscopic Modified Lothrop Procedure Using a Porcine Intestinal Submucosal Graft
Brief Title: Improvement of Outcomes in Draf III/Endoscopic Modified Lothrop Procedure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided to do a different clinical trial opportunity.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey D. Suh, Assistant Professor, Department of Head and Neck Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-001257
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Chronic Sinusitis; Frontal Sinusitis
Keywords: Chronic sinusitis; Frontal sinusitis; Skull base neoplasm
MeSH Terms: conditions — Frontal Sinusitis; Skull Base Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects within the control arm will undergo the Draf III/Endoscopic Modified Lothrop procedure to address their sinus disease. At the end of the procedure, no Cook Biodesign Porcine intestinal submucosal graft will be used to cover the operative site. Light nasal packing will be placed in the nasal cavity for hemostasis. No placebo will be utilized.
- Cook Biodesign (Experimental): Subjects within the experimental group will undergo the Draf III/Endoscopic Modified Lothrop procedure to address their sinus disease. At the end of the procedure, a small piece of Cook Biodesign porcine intestinal submucosal xenograft will be used to cover the exposed bone of the operative site along the frontal beak. It will be bolstered with light nasal packing to keep the graft in place during healing.
  Interventions: Device: Porcine Intestinal submucosal xenograft

INTERVENTIONS:
Device: Porcine Intestinal submucosal xenograft — Cook Biodesign ENT repair graft will be used in the experimental group to cover exposed bone in the sinonasal cavity as a result of the Draf III/endoscopic modified lothrop procedure.
  Other Names: Cook Biodesign ENT Repair
  Arms: Cook Biodesign

SUMMARY:
We propose a randomized, single-blinded, prospective trial in order to evaluate the efficacy of the Cook Biodesign ENT Repair graft in improving outcomes after the Draf III or Endoscopic Modified Lothrop procedure. The Cook Biodesign ENT Repair graft is a porcine intestinal submucosal xenograft which has been FDA approved for use as an adjunct to natural healing process in the sinonasal cavity. The Draf III or Endoscopic Modified Lothrop involved creating a large unified drainage pathway for refractory frontal sinusitis. After the procedure is completed, there is exposed bone along the frontal beak region which can become a nidus for inflammation, crusting and eventual scarring, leading to stenosis or even complete blockage of the frontal sinuses. The Cook Biodesign will be used to cover this exposed bone in order to potentially reduce the inflammation, crusting and scarring and possibly improve outcomes.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is an inflammatory disorder affecting the sinonasal mucosa. Chronic symptoms include facial pain and pressure, nasal airway obstruction, anosmia and nasal discharge (sometimes purulent), in addition to significant effects on overall quality of life. The cost of CRS is estimated to be approximately $4 billion per year and results in over 20 million physician visits per year. The frontal sinuses are paired paranasal sinuses housed superiorly and anteriorly in the frontal bone on each side, separated by an inter-sinus septum which is contiguous with the nasal septum. The frontal sinuses, like the other paranasal sinuses, can be affected in chronic rhinosinusitis, with inflammation of the frontal sinus outflow tract causing obstruction and subsequent symptoms. First line therapy involves medical therapy often with combination of antibiotics, nasal saline irrigation, topical and/or systemic corticosteroids, with endoscopic sinus surgical therapy reserved for patients with persistent symptoms after medical therapy.

Surgical therapy of the frontal sinus is the most technically demanding aspect of endoscopic sinus surgery, and due to this, surgical dissection of the frontal sinuses has been discouraged in the past. Otolaryngology textbooks also emphasize that chronic frontal sinus disease may be related to unnecessary instrumentation of the frontal recess. With recent advances in endoscopic sinus surgery and the advent of balloon sinusotomy, the rate of frontal sinus surgery has more than doubled from 2000 to 2009.

Primary frontal sinus surgery can be approached with balloon dilation or by endoscopic sinusotomy. Endoscopic sinusotomy of the frontal sinus involves increasing the size of the frontal recess with anterior ethmoidectomy and removal of the agger nasi cell anteriorly, and any frontal cells that may be present. Frontal sinus surgery is effective, as evidenced by a recent study analyzing long-term results after primary frontal sinus surgery showing a patency rate of 92% in a nearly 2-year average follow up period.

Refractory frontal sinusitis can be addressed surgically through external or 'extended' endonasal approaches. Historically, external approaches were first utilized, with introduction of osteoplastic flap techniques by Brieger in the 1890s. Lothrop introduced the Lothrop Procedure in 1914 which required an osteoplastic flap with removal of the frontal sinus floor and intersinus septum along with the upper aspect of the nasal septum to create a unified drainage pathway for the frontal sinuses. In the 1950s, Montgomery popularized the frontal sinus obliteration through osteoplastic flap approach leaving the frontal sinuses permanently non-functional through obliteration with fat or other materials. Though these external approaches often had high success rates, they require extensive dissection and are associated with a high morbidity and complication rate upwards of 20%. These complications included dural exposure, dural laceration with cerebrospinal fluid leak, orbital injury, forehead numbness, osteomyelitis and mucocele formation.

In 1991, Wolfgang Draf described an endoscopic approach to create a common drainage pathway akin to the Lothrop procedure which is now called the Endoscopic Modified Lothrop (EMLP) or Draf III procedure. Currently, the EMLP provides an endoscopic alternative for persistent frontal sinus disease after initial frontal sinusotomy, prior to consideration of frontal sinus obliteration through an osteoplastic flap approach. The EMLP involves drilling out the frontal sinus ostia on both sides and combining them through a superior septectomy, creating a large common drainage pathway for the two frontal sinuses. The EMLP offers reduced morbidity, shorter hospital stay, improved cosmetics, reduced blood loss and preservation of a functional frontal sinus. One meta-analysis study of 18 observational studies showed a restenosis rate of 19% and an overall failure rate of 13.9% (with failure defined as requiring revision surgery), with failure rates ranging from 0-33%. Restenosis of the frontal sinus ostium after EMLP is often attributed to a combination of scarring, adhesions or neo-osteogenesis, which occurs secondary to exposed bone after the surgical procedure. The exposed osteitic bone is believed to act as a source for inflammation and osteoblastic activity. Persistent mucosal disease has also been postulated as a contributor to postoperative stenosis after EMLP. Prevention of restenosis has been attempted with use of stents or medical therapy with topical application of mitomycin C and steroids with variable results.

Recent studies have attempted to address this issue by using mucosal grafts to cover the exposed frontal bone after EMLP. These studies describe using free or pedicled mucosal grafts from various sites in the nasal cavity to cover the bare bone exposed after EMLP drill out procedure. Two studies reported results using free mucosal grafts to cover the exposed bone and showed encouraging results, with patency rates 95% and 100%. Another study using a pedicled flap based off the anterior ethmoidal artery showed no restenosis in 4 patients. These studies utilize mucosa mostly from the nasal septum at the region of the superior septectomy which would otherwise be discarded, but they do also report use of inferior turbinate mucosa harvesting. Though minimal morbidity related to mucosal harvest was reported, any mucosal harvest from sites other than the operative site has the potential for creating additional postoperative morbidity. In addition, use of mucosa from a diseased mucosal cavity may not be optimal. Reducing rates of restenosis and failure in EMLP will allow for improved outcomes following this procedure and may prevent progression to more invasive and extensive surgical procedures.

This study will utilize a proprietary porcine intestinal submucosa graft Cook Biodesign™ ENT Repair graft to cover the exposed bone on the nasofrontal beak region following EMLP in order to evaluate its effects on mucosal healing and reduction of restenosis rates of the surgically augmented frontal sinus ostium after the Endoscopic Modified Lothrop Procedure. The Cook Biodesign™ ENT Repair for nasal mucosal replacement has been in use for sinonasal surgery since its Food and Drug Administration (FDA) approval in 2013. The Cook Biodesign™ ENT Repair graft is FDA approved for prescription use to "separate tissue or structures compromised by surgical trauma, help control minimal bleeding, and act as an adjunct to aid in the natural healing process. The device is indicated for use where an open wound dressing material is required in the nasal and/or sinus cavities following nasal and/or sinus surgery where separation of tissues or structures is desired."

The use of xenograft material in the method proposed in this submission has not been studied extensively. However, using free mucosal grafts or pedicled mucosal flaps after EMLP as previously discussed, have shown promise. The Cook Biodesign™ has been used preliminarily with patients in this proposed setting with good anecdotal results, including reduced crusting and good postoperative outcomes, however, its use has not yet been formally evaluated. The Cook Biodesign™ graft has several advantages over using native mucosal grafts: it is readily available and does not require harvest thus reducing operative times and potential morbidity from mucosa harvest sites, it is thinner than sinus mucosa and handled with ease, and it has tissue characteristics that promote wound healing. With the Cook Biodesign™, our hypothesis is that its use after EMLP surgery will allow for reduction of exposed bone in the sinonasal cavity and thus reduce inflammation, crusting and ultimately reduce restenosis and failure rates. Additionally, we hypothesize that reduction of crusting and inflammation will lead to improved patient reported symptom and quality of life scores on the Sinonasal Outcomes Test-22 (SNOT-22) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Any patient older than 18 years of age
* Frontal sinusitis refractory to previous surgical and/or medical therapy
* Patient with skull base neoplasm which requires Draf III or Endoscopic Modified Lothrop for exposure in excision of tumor

Exclusion Criteria:

* Previous Draf III or Endoscopic Modified Lothrop Procedure
* Allergy or objection to use of porcine-based graft material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Frontal sinus stenosis | 1 year
  Evaluate the size of the frontal sinus outflow tract over one year after surgery

SECONDARY OUTCOMES:
Number of postoperative debridements | 1 year
  Track the number of debridements required in the postoperative period
Need for further surgical intervention | 1 year
  Track if any further surgical procedures (in office or in operating room) that are required during postoperative period
Number of postoperative infections | 1 year
  Track the number of postoperative sinus infections, proven by culture, as well as the number of antibiotic courses required for treatment.
Lund Kennedy Endoscopy Score | 1 year
  Evaluation of the sinuses using nasal endoscopy and objective measurement using the validated Lund-Kennedy Endoscopy score
SNOT-22 score | 1 year
  Evaluation of patient quality of life using a validated questionnaire called the Sinonasal Outcome Test (SNOT) - 22.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Suh, MD, Principal Investigator — University of California Los Angeles, Department of Head and Neck Surgery
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pleis JR, Lucas JW. Summary health statistics for U.S. adults: National Health Interview Survey, 2007. Vital Health Stat 10. 2009 May;(240):1-159. PMID 19645319
- [Background] Naidoo Y, Wen D, Bassiouni A, Keen M, Wormald PJ. Long-term results after primary frontal sinus surgery. Int Forum Allergy Rhinol. 2012 May-Jun;2(3):185-90. doi: 10.1002/alr.21015. Epub 2012 Jan 17. PMID 22253224
- [Background] Pynnonen MA, Davis MM. Extent of sinus surgery, 2000 to 2009: a population-based study. Laryngoscope. 2014 Apr;124(4):820-5. doi: 10.1002/lary.24335. Epub 2013 Oct 2. PMID 23900802
- [Background] Anderson P, Sindwani R. Safety and efficacy of the endoscopic modified Lothrop procedure: a systematic review and meta-analysis. Laryngoscope. 2009 Sep;119(9):1828-33. doi: 10.1002/lary.20565. PMID 19554631
- [Background] Wormald PJ. Salvage frontal sinus surgery: the endoscopic modified Lothrop procedure. Laryngoscope. 2003 Feb;113(2):276-83. doi: 10.1097/00005537-200302000-00015. PMID 12567082
- [Background] Tran KN, Beule AG, Singal D, Wormald PJ. Frontal ostium restenosis after the endoscopic modified Lothrop procedure. Laryngoscope. 2007 Aug;117(8):1457-62. doi: 10.1097/MLG.0b013e31806865be. PMID 17585278
- [Background] Ye T, Hwang PH, Huang Z, Huang Q, Xian J, Li C, Zhou B. Frontal ostium neo-osteogenesis and patency after Draf III procedure: a computer-assisted study. Int Forum Allergy Rhinol. 2014 Sep;4(9):739-44. doi: 10.1002/alr.21357. Epub 2014 Jul 30. PMID 25079177
- [Background] AlQahtani A, Bignami M, Terranova P, Digilio E, Basilico F, Abdulrahman S, Castelnuovo P. Newly designed double-vascularized nasoseptal flap to prevent restenosis after endoscopic modified Lothrop procedure (Draf III): laboratory investigation. Eur Arch Otorhinolaryngol. 2014 Nov;271(11):2951-5. doi: 10.1007/s00405-014-2961-2. Epub 2014 Mar 8. PMID 24609647
- [Background] Conger BT Jr, Riley K, Woodworth BA. The Draf III mucosal grafting technique: a prospective study. Otolaryngol Head Neck Surg. 2012 Apr;146(4):664-8. doi: 10.1177/0194599811432423. Epub 2012 Jan 6. PMID 22228601
- [Background] Hildenbrand T, Wormald PJ, Weber RK. Endoscopic frontal sinus drainage Draf type III with mucosal transplants. Am J Rhinol Allergy. 2012 Mar-Apr;26(2):148-51. doi: 10.2500/ajra.2012.26.3731. PMID 22487293
- [Background] Seyedhadi S, Mojtaba MA, Shahin B, Hoseinali K. The Draf III septal flap technique: a preliminary report. Am J Otolaryngol. 2013 Sep-Oct;34(5):399-402. doi: 10.1016/j.amjoto.2013.01.019. Epub 2013 Feb 26. PMID 23452383
- [Background] Wei CC, Sama A. What is the evidence for the use of mucosal flaps in Draf III procedures? Curr Opin Otolaryngol Head Neck Surg. 2014 Feb;22(1):63-7. doi: 10.1097/MOO.0000000000000023. PMID 24335916